CLINICAL TRIAL: NCT05935462
Title: A Preliminary Study on the Demand and Design of Digital Learning Aids for Special Children With TRIZ and 3D Printing Technology
Brief Title: A Preliminary Study on Digital Learning Aids for Special Children With TRIZ and 3D Printing Technology
Status: Available | Type: Expanded Access
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: TMU-JIRB N202305081
Record Dates: First submitted 2023-06-23; First posted 2023-07-07 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-11

CONDITIONS: Digital Learning Aids for Special Children

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Combination Product: Digital Learning Aids — Recruitment is currently underway for special children undergoing outpatient early intervention. Among the recruited participants, five children between the ages of 6 and 9, who are receiving early intervention, were screened. After obtaining their consent to participate in this study, their basic information was recorded, including gender, age, education, diagnosis, Movement Assessment Battery for Children (MABC-2), Visual-Motor Integration (VMI) test, and Children's ABILHAND questionnaire for manual ability. Once the collection of basic information is completed, a trial of digital aids will be conducted, and a trial feedback questionnaire will be administered. The trial period will consist of a 20-minute session and 2-3 sessions (per week) of home (or therapy room) use.

SUMMARY:
During the transition phase from early intervention to primary education (4.5 years to 8.11 years), children with special needs may encounter difficulties in using digital learning media. The investigators intend to apply the TRIZ analysis method to enhance children's participation in learning. Additionally, the investigators plan to design a preliminary model of learning aids and conduct a trial.

DETAILED DESCRIPTION:
The design of digital learning aids for early childhood education for special children to participate in classroom learning is based on the principle of TRIZ analysis combined with the design of 3D printing technology to explore the needs and design of digital apparatus for early childhood education for special children to participate in classroom learning.

A exploratory study. Part 1: Analysis of Systematic Questionnaires. Thirty questionnaires were collected from users of learning devices based on the theoretical basis of ACCESS-FM.The results of the questionnaire are based on the theoretical concept analysis of TRIZ and are used for the preliminary design of learning aids.Part 2: Analysis of Assistive Device Trial. Five school-age children were recruited from the questionnaires for the preliminary design of learning aids. The results are collected for the digital platform performance (writing and typing tests), the ABILHAND-Kids, the Berry-Buktenica Developmental Test of Visual-Motor Integration, Motor Coordination, and the Children's Learning Devices. Motor Integration, Motor Coordination), the Movement Assessment Battery for Children for Children, Second Edition, the Quebec User Evaluation of Satisfaction with Assistive Technology; QUEST) and side effects.

Data Analysis: The performance and side effects of the digital platform operations before and after training were compared using Wilcoxon Signed Ranked Test. SPSS 20.0 was used and the level of statistically significant difference was set at Alpha<0.05.

ELIGIBILITY:
Inclusion Criteria:

Analysis of Systematic Questionnaires part

* the caregiver of a child with special needs in early care;
* the caregiver or child has trouble using electronic devices or needs;
* the child can cooperate with the full questionnaire;
* the child with special needs in early care attends school. Analysis of Assistive Device Trial part
* Special children aged 6 to 9 years who are currently receiving early intervention;
* Children who experience difficulties or have needs related to using electronic devices;
* Participants who are able to complete the trial sessions;
* Special children receiving early intervention who are attending school.

Exclusion Criteria:

Analysis of Systematic Questionnaires part

* The child is younger than 4.5 years old or older than 9 years old;
* The caregiver is unable to communicate and read in Chinese.

Analysis of Assistive Device Trial part

* Children younger than 6 years or older than 9 years of age;
* Children who are unable to recognize Zhuyin (Bopomofo) phonetic symbols.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

REFERENCES:
- [Result] Amaral DS, Duarte ALBP, Barros SS, Cavalcanti SV, Ranzolin A, Leite VMM, Dantas AT, Oliveira ASCRC, Santos PS, Silva JCA, Marques CDL. Assistive devices: an effective strategy in non-pharmacological treatment for hand osteoarthritis-randomized clinical trial. Rheumatol Int. 2018 Mar;38(3):343-351. doi: 10.1007/s00296-017-3892-1. Epub 2017 Nov 28. PMID 29185087
- [Result] Baronio G, Harran S, Signoroni A. A Critical Analysis of a Hand Orthosis Reverse Engineering and 3D Printing Process. Appl Bionics Biomech. 2016;2016:8347478. doi: 10.1155/2016/8347478. Epub 2016 Aug 9. PMID 27594781
- [Result] Funch A, Kruse NB, la Cour K, Peoples H, Waehrens EE, Brandt A. The association between having assistive devices and activities of daily living ability and health-related quality of life: An exploratory cross-sectional study among people with advanced cancer. Eur J Cancer Care (Engl). 2019 May;28(3):e13002. doi: 10.1111/ecc.13002. Epub 2019 Feb 10. PMID 30740805
- [Result] Keller M, Guebeli A, Thieringer F, Honigmann P. Overview of In-Hospital 3D Printing and Practical Applications in Hand Surgery. Biomed Res Int. 2021 Mar 26;2021:4650245. doi: 10.1155/2021/4650245. eCollection 2021. PMID 33855068
- [Result] Long TM, Woolverton M, Perry DF, Thomas MJ. Training needs of pediatric occupational therapists in assistive technology. Am J Occup Ther. 2007 May-Jun;61(3):345-54. doi: 10.5014/ajot.61.3.345. PMID 17569392
- [Result] Ma HI, Hwang WJ, Tsai PL, Hsu YW. The effect of eating utensil weight on functional arm movement in people with Parkinson's disease: a controlled clinical trial. Clin Rehabil. 2009 Dec;23(12):1086-92. doi: 10.1177/0269215509342334. PMID 19906764
- [Result] McDonald SS, Levine D, Richards J, Aguilar L. Effectiveness of adaptive silverware on range of motion of the hand. PeerJ. 2016 Feb 15;4:e1667. doi: 10.7717/peerj.1667. eCollection 2016. PMID 26893960
- [Result] Roda-Sales A, Vergara M, Sancho-Bru JL, Gracia-Ibanez V, Jarque-Bou NJ. Effect on hand kinematics when using assistive devices during activities of daily living. PeerJ. 2019 Oct 8;7:e7806. doi: 10.7717/peerj.7806. eCollection 2019. PMID 31608177
- [Result] Skymne C, Dahlin-Ivanoff S, Claesson L, Eklund K. Getting used to assistive devices: ambivalent experiences by frail elderly persons. Scand J Occup Ther. 2012 Mar;19(2):194-203. doi: 10.3109/11038128.2011.569757. Epub 2011 May 2. PMID 21534712